CLINICAL TRIAL: NCT07244848
Title: Effects of the Zinde Zihin Multidomain Lifestyle Program on Alzheimer's Disease Risk: A Two-Center Controlled Intervention Study
Brief Title: Zinde Zihin Program to Reduce Alzheimer's Disease Risk in Adults Aged 65 and Older
Acronym: ZZ-MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Ayse Sezer Balci, Assistant Professor, PhD, RN - Department of Public Health Nursing, Burdur Mehmet Akif Ersoy University, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAKU-ZINDEZIHIN-2025; Ethics Approval No: GO-2025/10 (Other: Burdur Mehmet Akif Ersoy University)
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Decline; Aging; Alzheimer Disease
Keywords: Alzheimer's Disease Risk; Cognitive Health; Aging; Multidomain Lifestyle Intervention; Older Adults
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Intervention Model Description:
  Participants are individually randomized into two parallel groups (intervention and control). The intervention group receives the Zinde Zihin multidomain lifestyle program, delivered in eight structured sessions over four weeks. The program includes cognitive stimulation, physical activity, nutrition education, psychosocial engagement, and sleep/stress management activities. Sessions are group-based and facilitated by a trained researcher. The control group receives routine nursing home activities without any additional structured intervention. Baseline and post-intervention assessments are administered to all participants. The model aims to examine changes in Alzheimer's Disease Risk Index scores and related lifestyle factors under a parallel assignment design.
Who Masked: Outcomes Assessor
Masking Description: Due to the behavioral nature of the intervention, participants and facilitators were aware of group assignments. However, data collection and statistical analysis were conducted by independent researchers who were blinded to group allocation to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinde Zihin (Fit Mind) Multidomain Lifestyle Intervention (Experimental): Participants in the intervention group received the eight-session Zinde Zihin (Fit Mind) multidomain lifestyle program, which combined cognitive training, moderate physical exercise, nutritional education, and psychosocial stimulation. Sessions were conducted twice weekly for four weeks in small group settings at nursing homes.
  Interventions: Behavioral: Zinde Zihin (Fit Mind) Multidomain Lifestyle Intervention
- Control Group - Routine Care (No Intervention): Participants assigned to the control group continued their usual daily activities and standard care routines in the nursing home. They did not receive any structured sessions of the Zinde Zihin (Fit Mind) program or other organized lifestyle interventions during the study period.

INTERVENTIONS:
Behavioral: Zinde Zihin (Fit Mind) Multidomain Lifestyle Intervention — The Zinde Zihin (Fit Mind) program is a culturally adapted multidomain lifestyle intervention developed to enhance cognitive health, emotional well-being, and daily functioning in older adults. The program combines four evidence-based components-cognitive training, physical activity, nutritional education, and psychosocial stimulation-delivered in eight 60-75-minute sessions over four weeks. Activities included memory and problem-solving games, balance and stretching exercises, discussions on brain-healthy diets, and group-based art, music, and storytelling exercises to strengthen social engagement and mental resilience.
  What distinguishes the Zinde Zihin program from other interventions is its cultural adaptation for Turkish older adults living in institutional settings. It integrates traditional Turkish music, storytelling, and collective art creation to increase emotional connection and sustainability. Sessions were held in small groups at nursing homes and facilitated by trained p
  Other Names: Fit Mind Program; Multidomain Lifestyle Intervention; Cognitive Health Promotion Program; Healthy Aging Behavioral Program
  Arms: Zinde Zihin (Fit Mind) Multidomain Lifestyle Intervention

SUMMARY:
This study aims to evaluate the feasibility and implementation of the Zinde Zihin ("Fit Mind") multidomain lifestyle program for older adults aged 65 years and older living in public nursing homes. The program includes cognitive activities, physical exercises, nutrition education, psychosocial engagement, sleep education, and stress-management components delivered in eight structured sessions over four weeks. The primary objective is to examine changes in Alzheimer's Disease Risk Index-Short Form (ANU-ADRI-SF) scores from baseline to post-intervention. Secondary objectives include assessing changes in cognitive activity engagement and affect-related lifestyle factors.

DETAILED DESCRIPTION:
The Zinde Zihin ("Fit Mind") Program is a multidomain lifestyle intervention designed to promote healthy cognitive aging among older adults. The intervention integrates cognitive training, physical activity, nutritional education, psychosocial engagement, and sleep/stress management techniques within a group-based framework. The program is delivered in eight structured sessions over four weeks, with each session lasting approximately 60-75 minutes.

Study Rationale Lifestyle factors such as cognitive stimulation, physical activity, sleep, and social engagement play an important role in cognitive health. Multidomain interventions involving these components may support healthy aging. This study was developed to examine the feasibility of such an intervention in Turkish nursing home settings.

Study Design This is an individually randomized, controlled pretest-posttest study conducted in two public nursing homes. Randomization is performed at the individual level after eligibility screening. The protocol follows CONSORT guidelines for individually randomized trials.

Participants Eligible participants are adults aged 65 years or older with a Mini-Mental State Examination (MMSE) score ≥23 who are able to communicate verbally and volunteer to participate. Exclusion criteria include diagnosed dementia, major psychiatric illness, severe sensory impairment preventing participation, or unwillingness to attend intervention sessions.

Intervention

Eight structured sessions are delivered to the intervention group:

* Orientation and baseline assessment
* Cognitive stimulation activities
* Emotional well-being and social interaction activities
* Physical activity and brain-health education
* Creative expression and art-based engagement
* Nutrition and brain-healthy dietary education
* Sleep education and relaxation techniques
* Reflection, feedback, and post-test assessment

The control group receives routine nursing home activities only.

Outcome Measures

Primary Outcome:

The Alzheimer's Disease Risk Index-Short Form (ANU-ADRI-SF), a self-report instrument assessing demographic, lifestyle, and medical factors associated with Alzheimer's disease risk. Scores are collected at baseline and at 4 weeks.

Secondary Outcomes:

Measures assessing cognitive activity participation and affect-related lifestyle factors, collected at baseline and 4 weeks.

Randomization and Allocation Concealment Participants are randomized using a computer-generated list stratified by institution. Allocation is concealed through sequentially numbered, opaque, sealed envelopes prepared by an independent researcher.

Blinding Due to the nature of the intervention, participants and facilitators cannot be blinded. Outcome assessors and data analysts remain blinded.

Ethics The study was approved by the Burdur Mehmet Akif Ersoy University Ethics Committee (GO 2025/1069). Written informed consent is obtained from all participants.

Data Collection and Timing Baseline and post-intervention assessments are administered individually by the researcher in a private room within the nursing homes.

Statistical Analysis Plan Descriptive statistics and statistical procedures appropriate to the data structure will be applied. Analyses will be conducted according to the predefined analysis plan.

ELIGIBILITY:
Inclusion Criteria:

Ages Eligible for Study:

65 Years to 80 Years (Older Adult)

Sexes Eligible for Study:

All

Accepts Healthy Volunteers:

Yes

Exclusion Criteria:

* Diagnosis of dementia or severe cognitive impairment.
* History of depression or major psychiatric disorder.
* Physical disability or medical condition prevents participation in exercise.
* Attendance in less than two-thirds of the planned intervention sessions.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in ANU-ADRI-SF Total Risk Score | Baseline (Week 0) to Post-intervention (Week 4)
  The Alzheimer's Disease Risk Index - Short Form (ANU-ADRI-SF; 45 items, 15 subscales) is a self-report instrument summing risk and protective factors; higher total scores indicate higher Alzheimer's disease risk. The primary endpoint is the change score (post - baseline). Negative values indicate risk reduction. Analyses will compare groups adjusting for cluster randomization (ICC).

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Sezer Balci, PhD, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Mehmet Akif Ersoy University Faculty of Health Science, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared because the dataset contains sensitive personal health information collected from older adults living in nursing homes. Only aggregate (group-level) data will be published in scientific journals upon request.